CLINICAL TRIAL: NCT06948487
Title: A Prospective, Multi-center, Observational Study on the Efficacy and Safety of FEXUCLUE Tab. In Patients With Acute or Chronic Gastritis
Brief Title: Efficacy and Safety of FEXUCLUE Tab. In Patients With Acute or Chronic Gastritis
Status: Recruiting | Type: Observational
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Other Study IDs: DW_FEX_DB_03
Record Dates: First submitted 2025-04-15; First posted 2025-04-29 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Gastritis
Keywords: Acute; Chronic
MeSH Terms: conditions — Gastritis; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fexuclue® Tab: Fexuclue® Tab Fexuclue® Tab Fexuprazan Hydrochloride 10mg

SUMMARY:
This study aims to evaluate the efficacy of Fexuclue tablets in improving gastrointestinal symptoms based on patient-reported outcomes (PROs), by comparing assessments before and after treatment.

DETAILED DESCRIPTION:
In this observational study, patient-reported data will be collected using an electronic application (e-PRO). The survey on subjective symptoms will be administered twice-once before and once after the administration of Fexuclue tablets. Additionally, a survey on medication convenience will be conducted once at 2 weeks (up to a maximum of 4 weeks) post-administration.

At the same time point (2 to 4 weeks after administration), patients will self-assess their overall improvement through the e-PRO application. Investigators will also evaluate final improvement based on clinical judgment in a real-world setting and record the outcome in the Case Report Form (CRF).

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects between the ages of 19 and 75 years at the time of obtaining written informed consent.
* Subjects who are scheduled to receive Fexuclu tablets (fexuprazan) in accordance with the approved indication.
* Subjects who present with at least one subjective symptom requiring medical treatment
* Subjects who are capable of understanding the information provided, have voluntarily decided to participate in this observational study, and have provided written informed consent for the use of their personal data.

Exclusion Criteria:

* Individuals who fall under any contraindications for the administration of Fexuclu tablets (fexuprazan) as specified in the approved labeling.
* Individuals who are deemed by the investigator (attending physician) to be inappropriate for participation in this observational study for any reason not otherwise specified.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The proportion of subjects with improved subjective symptoms at 2 to 4 weeks after Fexuclue tablet administration for gastritis will be assessed based on patient-reported outcomes. Referring to prior Phase 3 data, a 60% efficacy rate is assumed. Using G-Power 3.1.9.7 with a two-sided significance level of 0.05 and statistical power of 95%, the minimum sample size was calculated to be 10,434. Considering a 25% dropout rate, approximately 13,000 participants will be enrolled.
Sampling Method: Probability Sample
Enrollment: 12000 (Estimated)
Dates: Start 2025-06-17 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2027-06-03 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects with improvement in subjective symptoms | 2 weeks(up to 4 weeks)
  The proportion of subjects with improvement in subjective symptoms at Week 2 (up to Week 4) compared to baseline.

SECONDARY OUTCOMES:
Change from baseline in the mean frequency scores of individual subjective symptoms assessed at each time point using a 5-point scale ranging from 0 (not at all) to 4 (daily) | 2 weeks(up to 4 weeks)
  Change from baseline in the mean frequency scores of individual subjective symptoms assessed at each time point using a 5-point scale ranging from 0 (not at all) to 4 (daily) at 2 weeks(up to 4 weeks)
Change from baseline in the mean severity scores of individual subjective symptoms assessed at each time point using a 5-point scale ranging from 0 (not at all) to 4 (very severe) | 2 weeks(up to 4 weeks)
  Change from baseline in the mean severity scores of individual subjective symptoms assessed at each time point using a 5-point scale ranging from 0 (not at all) to 4 (very severe) at 2 weeks(up to 4 weeks)
Disappearance rate of subjective symptoms | 2 weeks(up to 4 weeks)
  Disappearance rate of subjective symptoms at 2 weeks(up to 4 weeks)
Overall improvement assessed at each time point by both the subject and the investigator using the Final Improvement Assessment, which consists of a 5-point scale ranging from 'fully recovered' to 'worsened' | 2 weeks(up to 4 weeks)
  Overall improvement assessed at each time point by both the subject and the investigator using the Final Improvement Assessment, which consists of a 5-point scale ranging from 'fully recovered' to 'worsened' at 2 weeks(up to 4 weeks)
Patient-reported satisfaction with medication intake convenience assessed at Week 2 (up to Week 4) compared to baseline, using a 5-point scale ranging from 'very convenient' to 'very inconvenient' | 2 weeks(up to 4 weeks)
  Patient-reported satisfaction with medication intake convenience assessed at Week 2 (up to Week 4) compared to baseline, using a 5-point scale ranging from 'very convenient' to 'very inconvenient' at 2 weeks(up to 4 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Jingun Kim, Dr., Principal Investigator — Masong Kim Internal Medicine Clinic
Locations (1):
- Masong Kim Internal Medicine Clinic, Seoul, South Korea